CLINICAL TRIAL: NCT00835991
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Glyburide/Metformin 5 mg/500 mg Film-Coated Tablets and Glucovance® 5 mg/500 mg Film-Coated Tablets in Healthy Subjects Under Fed Conditions
Brief Title: Glyburide/Metformin 5 mg/500 mg Film-Coated Tablets, Fed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02350
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Glyburide; Metformin; Glucovance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyburide Metformin (Experimental): Glyburide Metformin 5/500 Film-Coated Tablet (test) dosed in first period followed by Glucovance® 5/500 mg Tablet (reference) dosed in second period
  Interventions: Drug: Glyburide/Metformin 5 mg/500 mg Tablets
- Glucovance® (Active Comparator): Glucovance® 5/500 mg Tablet (reference) dosed in first period followed by Glyburide Metformin 5/500 mg Film-Coated Tablet (test) dosed in second period
  Interventions: Drug: Glucovance® 5 mg/500 mg Tablets

INTERVENTIONS:
Drug: Glyburide/Metformin 5 mg/500 mg Tablets — 1 x 5 mg/500 mg, single-dose fed
  Arms: Glyburide Metformin
Drug: Glucovance® 5 mg/500 mg Tablets — 1 x 5 mg/500 mg, single-dose fed
  Arms: Glucovance®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of Glyburide/Metformin 5 mg/500 mg film-coated tablets (test) versus Glucovance® (reference) administered as 1 x 5 mg/500 mg film-coated tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age and older.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* Subjects with BMI less than or equal to 30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* History of allergic reactions to glyburide or to metformin or other related drugs (e.g. chlorpropamide, gliclazide, tolbutamide, furosemide, sulfamethoxazole, sulfadiazine and sulfisoxazole).
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* History or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication except for topical products without systemic absorption.
* Positive alcohol breath test at screening. subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Intolerance to venipuncture.
* Any food allergy, intolerance, restriction, or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows: less than 300 mL of whole blood within 30 days or; 300 mL to 500 mL of whole blood within 45 days or; more than 500 mL of whole blood within 56 days.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* History of metabolic acidosis, congestive heart failure and myocardial infarction.
* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).
* Female subjects of childbearing potential who have had unprotected sexual intercourse with any non-steril male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. The acceptable methods of contraception are:

  1. Condom + spermicide
  2. Diaphragm + spermicide
  3. Intrauterine contraceptive device (placed at least 4 weeks prior to study drug administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Glyburide Metformin (Test) First: Glyburide Metformin 5/500 Film-Coated Tablet (test) dosed in first period followed by Glucovance® 5/500 mg Tablet (reference) dosed in second period
- Glucovance® (Reference) First: Glucovance® 5/500 mg Tablet (reference) dosed in first period followed by Glyburide Metformin 5/500 mg Film-Coated Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Glyburide Metformin (Test) First | Glucovance® (Reference) First
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout
Arm/Group | Glyburide Metformin (Test) First | Glucovance® (Reference) First
Started | 30 | 29
Completed | 27 | 26
Not Completed | 3 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1
Period: Second Intervention
Arm/Group | Glyburide Metformin (Test) First | Glucovance® (Reference) First
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glyburide Metformin (Test) First | Glucovance® (Reference) First | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 24 | 27 | 51
  American Hispanic | 4 | 2 | 6
  Black | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration) - Glyburide
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Glyburide Metformin: Glyburide Metformin 5/500 Film-Coated Tablet (test) dosed in either period
- Glucovance®: Glucovance® 5/500 mg Tablet (reference) dosed in either period
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng/mL | 190.17 (68.08) | 166.48 (59.87)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 114.05, 90% CI [107.26 to 121.27] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Glyburide
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng*h/mL | 970.22 (328.93) | 977.28 (402.74)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 100.63, 90% CI [97.59 to 103.76] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)] - Glyburide
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng*h/mL | 942.94 (316.17) | 943.45 (388.26)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 101.36, 90% CI [98.32 to 104.48] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Primary Outcome: Cmax (Maximum Observed Concentration) - Metformin
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng/mL | 755.10 (195.97) | 766.30 (210.22)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 99.05, 90% CI [94.31 to 104.02] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

5. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Metformin
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng*h/mL | 6308.12 (1662.69) | 6552.79 (1833.42)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.55, 90% CI [93.85 to 99.32] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

6. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)] - Metformin
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glyburide Metformin | Glucovance®
Number analyzed (Participants) | 53 | 53
ng*h/mL | 6203.57 (1656.57) | 6448.34 (1814.06)
Statistical Analysis 1: Comparison: Glyburide Metformin vs Glucovance®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.44, 90% CI [93.71 to 99.25] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.